CLINICAL TRIAL: NCT01566266
Title: Gut Flora and Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: METC 12-3-011
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Hypercholesterolemia
Keywords: gut flora; antibiotics; lipid metabolism; LDL cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin (Experimental)
  Interventions: Drug: Amoxicillin
- Placebo capsules (Placebo Comparator)
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Amoxicillin — 2 capsules of 250mg, 3 times per day during 1 week
  Arms: Amoxicillin
Drug: Placebo capsule — 2 capsules of 250mg, 3 times per day during 1 week
  Arms: Placebo capsules

SUMMARY:
It is well known that metabolic responses to diet and drugs are affected by genetic and environmental factors. Still, a large part of differences in responses between individuals remains unexplained. To increase our understanding of individual differences, more and more attention is paid to the role of intestinal microbiota. Not only energy and glucose may be related to the microbiota, but also lipid metabolism. This is not surprising as lipid metabolism, glucose metabolism, and obesity are closely linked.

There is substantial evidence from in particular animal studies that the gut microbiota is related to lipid and lipoprotein metabolism. However, there is less evidence to what extent modulation of the gut microbiota changes lipid and lipoprotein metabolism in humans.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18-70 years
* serum total cholesterol: 5-8mmol/L

Exclusion Criteria:

* serum triacylglycerol > 3.0mmol/L
* use of oral anticonceptives
* pregnant or breastfeeding women
* kidney insufficiencies
* unstable body weight
* allergy to antibiotics
* treatment with cholesterol-lowering drugs
* use of medication or a medically prescribed diet
* active cardiovascular disease
* abuse of drugs
* more than 21 alcohol consumptions per week for men and 14 consumptions for women
* use of an investigational product within the previous 30 days
* not willing to stop the consumption of products rich in plant stanol or sterol esters 3 weeks before start of the study
* use of gastric acid inhibitors, laxantia, prebiotica, probiotica and antibiotica for at least one month before the start of the study and during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol | Measure change between day 1 and day 8

SECONDARY OUTCOMES:
Lipid metabolism | Measure change between day 1 and day 8 (HDL-cholesterol, triglycerides)
Glucose metabolism | Measure change between day 1 and day 8

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Mensink, Prof. Dr. Ir., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands